CLINICAL TRIAL: NCT00426504
Title: Helical Tomotherapy Intensity Modulated Radiotherapy:A Phase I/II Pilot Study to Determine the Toxicity Profile, Pattern of Failures and Quality of Life of Patients With Squamous Cell Carcinoma of the Head and Neck
Brief Title: Radiation Therapy Using Helical Tomotherapy IMRT for Head and Neck Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005781-01H; OTT 05-06 (Other: OHRI)
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2020-07-30 (Actual); Status verified 2020-03

CONDITIONS: Cancer
Keywords: Head,; Neck,; Cancer,; Tomotherapy,; IMRT,
MeSH Terms: conditions — Neoplasms | interventions — Radiotherapy

ARMS (1):
- radiotherapy (Experimental): Helical Tomotherapy Intensity Modulated Radiotherapy (HT-IMRT) with the intend of delivering radical radiotherapy to a dose of 66-70 Gy to involved areas and at least 50 Gy to un-involved sites to be treated prophylactically.
  Interventions: Procedure: Radiotherapy

INTERVENTIONS:
Procedure: Radiotherapy — Helical Tomotherapy Intensity Modulated Radiotherapy (HT-IMRT) with the intend of delivering radical radiotherapy to a dose of 66-70 Gy to involved areas and at least 50 Gy to un-involved sites to be treated prophylactically.
  Other Names: Helical tomotherapy IMRT

SUMMARY:
Historically, patients with stage III and IV head and neck cancer have been treated with surgery and/or radiation therapy. Based on the results of recent clinical trials, in patients not able to undergo surgery, chemotherapy with radiation therapy has been adopted as the current standard of care. The chemo-radiation approach, however, entails a significant increase in treatment-related toxicity, limiting the extent to which this treatment can be offered to patients. In this trial, the ability of a new form of radiation therapy delivery called IMRT will be evaluated for its ability to reduce the amount of radiation-induced toxicity.

DETAILED DESCRIPTION:
The mechanisms of action to explain the radiation-induced toxic effects resulting from the more aggressive radiation therapy treatments of head and neck cancer include the additive and synergistic increase in mucositis from the combination of chemotherapy and radiotherapy. The severe toxicity associated with more aggressive radiation therapy treatments for locoregional head and neck cancer limits the extent to which these treatments can be offered since many patients present with nutritional deficiencies and consequent general debility. Intensity Modulated Radiotherapy (IMRT) is a technology has the potential for exquisite dose painting and structuring in such a manner that it can permit exclusion of normal tissues and sensitive structures from the high dose radiation volume without compromising primary tumor or nodal target coverage. In this phase I/II feasibility trial, radical radiotherapy will be delivered using Helical Tomotherapy Intensity Modulated Radiotherapy (HT-IMRT) to a dose of 66-70 Gy to involved areas and to at least 50 Gy to un-involved sites, treated prophylactically. It is hypothesized that the pattern of failure and toxicity profiles of patients treated with helical tomotherapy will demonstrate the greater efficacy of helical tomotherapy, as compared with conventional radiotherapy, in the treatment of cancers of the head and neck.

ELIGIBILITY:
Inclusion Criteria:

1. Stage II, III or IV non-metastatic histologically confirmed carcinoma of the head and neck region (Oral cavity, pharynx or larynx).
2. Treatment with radical radiotherapy with or without chemotherapy
3. Patients in whom definitive radiotherapy with or without planned neck dissection is the selected curative treatment
4. ECOG performance status of 0, 1 or 2

Exclusion Criteria:

1. Previous radiotherapy to head and neck mucosa
2. Patients with disabling co-morbid conditions, which do not permit effective immobilization
3. Patients with severe trismus, which disallow effective assessment
4. Patients in whom it is deemed necessary to commence enteric nutrition prior to the start of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2006-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
1) To determine the toxicity profile of patients with head and neck cancer treated with helical tomotherapy-IMRT | weekly
  MEASURING MUCOSITIS

SECONDARY OUTCOMES:
1) To compare the dose distributions generated by HT-IMRT with those generated using three-dimensional conformal radiation, 2) To determine the pattern of relapse in the primary site and neck within the first 2 years following treatment, | 1-once 2- 6 monthly
  comparing dose distribution

CONTACTS AND LOCATIONS:
Overall Officials: Samy El-Sayed, MD, Study Chair — OHRI
Locations (1):
- The Ottawa Hospital Regional Cancer Centre, Ottawa, Ontario, Canada